CLINICAL TRIAL: NCT03816072
Title: Simultaneous Quantification of Dynamic and Static Cerebral Autoregulation (CA) at Different Steady-state Mean Blood Pressures Under Anaesthesia.
Brief Title: Quantification of Dynamic and Static Cerebral Autoregulation (CA) Under Anaesthesia
Acronym: SAMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Niek Sperna Weiland, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: METC 2018_230
Record Dates: First submitted 2019-01-21; First posted 2019-01-25 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Cerebrovascular Circulation
MeSH Terms: interventions — Respiration, Artificial; Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: Patients receive either propofol or sevoflurane to maintain anaesthesia. Both treatment groups receive the same phenylephrine and mechanical ventilation regimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): ASA-I/II patients undergoing elective, non-cardiothoracic surgery with intravenous anaesthesia (propofol).
  Interventions: Drug: Phenylephrine infusion; Other: Mechanical ventilation; Drug: Propofol
- Sevoflurane (Active Comparator): ASA-I/II patients undergoing elective, non-cardiothoracic surgery with inhalational anaesthesia (sevoflurane).
  Interventions: Drug: Phenylephrine infusion; Other: Mechanical ventilation; Drug: Sevoflurane

INTERVENTIONS:
Drug: Phenylephrine infusion — Correction of anesthesia induced hypotension with phenylephrine to obtain sCA and dCA measurements at 60, 70, 80, 90 and 100 mmHg mean blood pressure. This is achieved by stepwise increases in phenylephrine infusion dose.
Other: Mechanical ventilation — Patientes are mechanically ventilated at 6 bpm to obtain low frequency blood pressure oscillations (~0.1 Hz).
Drug: Propofol — Propofol
  Arms: Propofol
Drug: Sevoflurane — Sevoflurane
  Arms: Sevoflurane

SUMMARY:
Cerebral autoregulation (CA) is the mechanism by which the brain vasculature maintains constancy of cerebral blood flow (CBF). Reliable direct measurements of CBF at different blood pressure levels are difficult because they are invasive and time-consuming. This type of measurement to quantify CA is generally referred to as static cerebral autoregulation (sCA). Alternatively, it is possible to measure CA indirectly from blood pressure oscillations. Dynamic cerebral autoregulation (dCA) measures how quickly the cerebral vessels react to a change in blood pressure to normalize CBF. Since the introduction of transcranial Doppler ultrasound (TCD), it has become possible to estimate CBF velocity relatively easy, which in turn correlates well with CBF changes. This method is widely used to quantify dCA. However, it is not clear how sCA correlates with dCA over a range of physiologic mean blood pressure (MBP). It is important to compare different methods of assessing CA, because impaired CA may result in increased risk of perioperative complications such as stroke. In this study, the investigators were interested in establishing the relationship between sCA and dCA during surgery under general anesthesia. The investigators aim to compare these methods during propofol and sevoflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA-I or ASA-II, willing and able to give written informed consent, scheduled for elective, non-cardiothoracic surgery under general anaesthesia and age 18 years and above.

Exclusion Criteria:

* Patient related

  * Unable/ unwilling to participate
  * ASA-III or higher
  * Age < 18 years
  * History of: uncontrolled hypertension, diabetes, Parkinson's disease, uncontrolled cardiac arrhythmia, Pure autonomic failure (formerly called idiopathic orthostatic hypotension), Multiple system atrophy with autonomic failure (formerly called Shy-Drager syndrome), Addison's disease and hypopituitarism, pheochromocytoma, peripheral autonomic neuropathy (e.g., amyloid neuropathy, idiopathic autonomic neuropathy), known cardiomyopathy, extreme left ventricle hypertrophy or ejection fraction < 30%, proven or suspected allergy for any of the medication used during induction of anaesthesia, malignant hyperthermia.
  * Unability to record transcranial Doppler ultrasound due to anatomical variance (~5% of population)
  * Contra-indications for intravenous or inhalational anaesthesia.
  * Contra-indications for phenylephrine: severe hypertension, peripheral vascular illness, severe hyperthyroidism
  * Simultaneous use of MAO-inhibitors, dopaminergic or vasoconstrictor ergot alkaloids (bromocriptine, cabergoline, pergolide, ergotamine, methylergometrine, methysergide), linezolid, tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitors, digoxin, quinidine, oxytocin.
* Surgery related

  * Day case surgery
  * Laparoscopy with CO2 insufflation
  * Extreme positioning during surgery (head-down/up tilt, lateral decubitus position, prone)
  * Surgery < 60 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Changes in dCA after several MBP-increasing steps. | Intraoperatively
Differences in dCA between sevoflurane and propofol at different steady-state MBP's. | Intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Hermanides, Dr., Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van den Dool REC, Sperna Weiland NH, Schenk J, Kho E, Veelo DP, van der Ster BJP, Immink RV. Dynamic cerebral autoregulation during step-wise increases in blood pressure during anaesthesia: A nonrandomised interventional trial. Eur J Anaesthesiol. 2023 Jun 1;40(6):407-417. doi: 10.1097/EJA.0000000000001798. Epub 2023 Feb 6. PMID 36655712